CLINICAL TRIAL: NCT05290181
Title: The Effect of Pilates Exercise and Whatsapp Text-Based Support Program on Premenstrual Syndrome (PMS) Symptoms: A Randomized Controlled Study
Brief Title: The Effect of Pilates Exercise and Whatsapp Text-Based Support Program on Premenstrual Syndrome (PMS) Symptoms
Acronym: PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ayca Balmumcu, Principal Investigator, Women's health and obstetrics nursing, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ABalmumcu
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Premenstrual Syndrome; Physical Exercise; Women's Health
Keywords: Premenstrual Syndrome; Pilates exercises; Text message; women's health
MeSH Terms: conditions — Premenstrual Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: 68 female students with PMS who met the inclusion criteria will be divided into groups using a simple random method. There will be 34 female students in the intervention group and 34 female students in the control group.In order to prevent interaction between the intervention and control group students in the randomization, the places where the students stay (home, dormitory rooms) will be taken into account. A support program including pilates exercises and sending text messages will be applied to the students in the intervention group for 8 weeks. Online pilates exercises will be done 2 days a week and individual short messages will be sent to their smartphones via the Whatsapp application 3 days a week.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise and whatsapp text message group (Experimental): A support program including pilates exercises and sending text messages will be applied to the students in the intervention group for 8 weeks. Online pilates exercises will be done 2 days a week and individual short messages will be sent to their smartphones via the Whatsapp application 3 days a week. Participants will be provided with Pre Pilates exercises, Pilates Mat Program: Beginner Level, Pilates Mat Program: Intermediate Level, Pilates Mat Program: Advanced level exercises. The exercises will be done online in the presence of a research physiotherapist with The Australian Physiotherapy & Pilates InstituteMatwork Level 1 (APPI) certificate.
  Interventions: Other: A support program with pilates exercise and whatsapp text message
- Control group (No Intervention): No intervention will be made in the control group.

INTERVENTIONS:
Other: A support program with pilates exercise and whatsapp text message — Female students in the intervention group will be given online pilates exercises 2 days a week for 8 weeks. Pre Pilates exercises, Pilates Mat Program: Beginner Level, Pilates Mat Program: Intermediate Level, Pilates Mat Program: Advanced level exercises will be provided. The exercises will be performed in the company of a research physiotherapist who has The Australian Physiotherapy & Pilates InstituteMatwork Level 1 (APPI) certificate. 3 days a week, individual short messages will be sent to the smartphones of female students via the Whatsapp application. General information about PMS will be sent in the first week, and motivational messages about lifestyle will be sent in the following weeks. Short message contents will be prepared by researchers in line with the literature and expert opinion will be taken. When the support program ends, PMSS will be applied to female students in the intervention group.
  Arms: Pilates exercise and whatsapp text message group

SUMMARY:
The aim of this study is to evaluate the effect of Pilates exercise and Whatsapp text message-based support program on PMS symptoms experienced by university female students.

DETAILED DESCRIPTION:
In this study, it will be answered whether the Pilates exercise and the support program based on Whatsapp text messages have an effect on the PMS symptoms experienced by university female students. Demographic information of the participants will be collected with the Personal Information form. The personal information form is a form prepared by the researchers with the support of the literature, consisting of 21 questions aiming to obtain information about the socio-demographic characteristics, menstrual characteristics, and lifestyle behaviors of the students. PMS symptoms will be evaluated with the Premenstrual Syndrome Scale. First of all, the premenstrual syndrome scale will be applied by trying to reach all 380 female students studying at the school. Afterward, 68 students with PMS who meet the inclusion criteria will be divided into 34 intervention and 34 control groups by simple randomization. In order to prevent interaction between the intervention and control group students in the randomization, the places where the students stay (home, dormitory rooms) will be taken into account. A support program including pilates exercise and WhatsApp text messages will be applied to the initiative group for 8 weeks. No attempt will be made on the control group.

ELIGIBILITY:
Inclusion Criteria:

* Having regular menstrual cycles (intervals of 21-35 days, lasting 3-10 days),
* Body mass index of 18.5-24.9 kg/m. to be between
* Absence of chronic disease,
* Absence of a hormonal disease such as polycystic ovary syndrome,
* Using smart mobile phone
* Not using oral contraceptives or antidepressants.

Exclusion Criteria:

* - Having a chronic or physical illness that prevents Pilates.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Premenstrual syndrome scale (PMSS) | Baseline
  The premenstrual syndrome scale (PMSS) aims to measure the severity of symptoms. The scale consists of 44 items in 5-point Likert type. The Cronbach's alpha value of the scale was determined as 0.75. As stated in the PMSS directive, while filling out the scale, the participants should mark according to the symptoms they felt one week before the period. In scoring the scale, the "Never" option is 1 point, the "Very little" option is 2 points, the "Sometimes" option is 3 points, the "Frequently" option is 4 points, and the "Constantly" option is evaluated. as 5 points. While evaluating the PMSS results, the presence of PMS is evaluated according to the condition of passing 50% of the highest score that can be obtained from the total and subscale scores. The highest possible score for the total score is 220, 50% of which is 110. A score above 110 points on the scale indicates the presence of PMS.

SECONDARY OUTCOMES:
Premenstrual syndrome scale (PMSS) | Immediately after the 8-week support intervention program
  The premenstrual syndrome scale (PMSS) aims to measure the severity of symptoms. The scale consists of 44 items in 5-point Likert type. The Cronbach's alpha value of the scale was determined as 0.75. As stated in the PMSS directive, while filling out the scale, the participants should mark according to the symptoms they felt one week before the period. In scoring the scale, the "Never" option is 1 point, the "Very little" option is 2 points, the "Sometimes" option is 3 points, the "Frequently" option is 4 points, and the "Constantly" option is evaluated. as 5 points. While evaluating the PMSS results, the presence of PMS is evaluated according to the condition of passing 50% of the highest score that can be obtained from the total and subscale scores. The highest possible score for the total score is 220, 50% of which is 110. A score above 110 points on the scale indicates the presence of PMS.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Balmumcu, PhD, Study Director — Aydin Adnan Menderes University
Locations (1):
- Aydin Adnan Menderes University, Aydin, Söke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No